CLINICAL TRIAL: NCT06468774
Title: Intestinal Ischemia Biomarker and Quality of Life of the Patients With Chronic Mesenteric Ischemia and Median Arcuate Ligament Syndrome
Brief Title: Intestinal Ischemia Biomarker in Patients With Chronic Mesenteric Ischemia
Status: Recruiting | Type: Observational
Sponsor: Oslo University Hospital (Other)
Responsible Party: Principal Investigator, Syed Sajid Hussain Kazmi, Principal Investigator, Oslo University Hospital
Other Study IDs: 607155
Record Dates: First submitted 2024-06-12; First posted 2024-06-21 (Actual); Last update posted 2025-07-30 (Actual); Status verified 2025-07

CONDITIONS: Chronic Mesenteric Ischemia; Median Arcuate Ligament Syndrome; Crohn Disease; Cholelithiasis
Keywords: Intestinal ishchemia biomarker; alpha GST; MALS; Chronic mesenteric ischemia
MeSH Terms: conditions — Median Arcuate Ligament Syndrome; Crohn Disease; Cholelithiasis | interventions — Laparoscopy; Angioplasty

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — plasma Alpha glutathione S transferase (Alpha GST)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (6):
- Median arcuate ligament syndrome (MALS): Patients with MALS Scheduled for laparoskopic decompression.
  Interventions: Procedure: Laparoscopic surgery
- Chronic mesenteric ischemia (CMI): Patients with CMI caused by atherosclerotic stenosis or occlusion of celiac artery, superior mesenteric artery ( one or both arteries ), and scheduled treatment with either PTA/stent or mesenteric bypass.
  Interventions: Procedure: Laparoscopic surgery
- Morbus Crohn intestine: Patients with diagnosed Mb Crohn of intestine who does not have CMI or MALS excluded with duplex ultrasound.
- Cholilithiasis: Patients with diagnosed Cholilithiasis who is scheduled for operative chelecystectomy and does not have CMI or MALS, excluded with the help of duplex ultrasound.
- Blood donor (Young): Healthy blood donor with a median age of 45 years, who does not have symptoms of mesenteric ischemia or MALS and has excluded these two conditions with the help of duplex ultrasound.
- Blood donor (Old): Healthy blood donor with a median age of 70 years, who does not have symptoms of mesenteric ischemia or MALS and has excluded these two conditions with the help of duplex ultrasound.

INTERVENTIONS:
Procedure: Laparoscopic surgery — The patients in the MALS group will be treated through transperitoneal ventral approach for the laparoscopic release of the celiac artery. Median arcuate ligament and any muscle or nerve tissue crossing the cranial surface of the celiac artery will be divided to release the celiac artery from compression.
  In the patients with CMI open antegrade or retrograde bypass to celiac artery or superior mesenteric artery or both will be performed.
  For operative treatment will be performed in general anaethesia whereas the endovacular treatment with PTA with stent for CMI will be performed in local anaethesia.
  Other Names: Percutaneous transluminal angioplasty (PTA) with stent; Open mesenteric bypass
  Groups: Chronic mesenteric ischemia (CMI); Median arcuate ligament syndrome (MALS)

SUMMARY:
Plasma Alpha glutathione S transferase (Alpha GST) has been previously demonstrated to be raised in patients with chronic mesenteric ischemia (CMI) caused by atherosclerosis and in patients with median arcuate ligament syndrome (MALS). Raised plasma level of Alpha GST has been demonstrated to decrease or normalize after surgical treatment of patients with CMI and MALS as compared with healthy individuals.

This study compares the plasma Alpha GST in patients with CMI and MALS with those with 1-Morbus Crohn, 2-Gallstone disease, and age-matched healthy individuals.

Besides, changes in the health-related quality of life (QoL) will be investigated in the study individuals.

DETAILED DESCRIPTION:
Patients with CMI and MALS usually complain of postprandial abdominal pain, changes in food intake pattern, and weight loss. These symptoms are often shared with many other more common diseases. Therefore, the diagnosis of CMI, and especially MALS, is often an exclusion diagnosis. To this date, no biomarker of intestinal ischemia with sufficient sensitivity and specificity has been identified for routine clinical use.

In a previous study, raised levels of plasma Alpha glutathione S transferase (Alpha GST) (7.8 ng/mL) in patients with CMI caused by atherosclerosis and in the patients with MALS (8.4 ng/mL). The raised plasma level of Alpha GST has been demonstrated to decrease or normalize after surgical improvement of the intestinal circulation in patients with CMI and MALS as compared with healthy individuals (3.3 ng/mL). However, the study was not appropriately powered and did not include a control group with similar clinical symptoms as in the patients with CMI and MALS.

This study will compare the plasma Alpha GST levels in patients with CMI (n=30) and MALS (n=30) with 1-Morbus Crohn (n=30), 2-Gallstone disease (n=30), and age-matched healthy individuals (n=60).

The CMI and MALS patients diagnosed with CTA and duplex ultrasound and scheduled to have either endovascular (PTA or stent) or open surgery (mesenteric bypass ) treatment will be included in this study.

Duplex ultrasound will be used to exclude CMI and MALS in the individuals in the control groups. After inclusion in the study, venous blood samples will be taken to exclude renal failure and liver disease. The blood samples will be repeated within 3 months. The blood samples will be centrifuged and stored at -70 degrees until analyzed in batches with the ELISA technique. Participants in the control groups will be examined with duplex ultrasound at the time of inclusion in the study and agian at three months.

In the patient groups, i.e., CMI and MALS, the venous blood samples will be obtained before and 3 months after the treatment. The blood samples will be centrifuged and stored at -70 degrees until analyzed in batches with the ELISA technique.

The plasma levels of Alpha GST will be compared beside receiver operating characteristic curves (ROC), and the area under the curve(AUC) will be calculated.

In addition to Alpha GST, the plasma of the study individuals will also be tested for other potential markers of intestinal ischemia, i.e., intestinal fatty acid binding protein (i-FABP), citrulline, and ischemia-modified albumin (IMA).

The study will also follow the patients participating in the study for clinical changes in symptoms. In addition, patient demographics, comorbidities, treatment demographics, and complications of the treatment will be registered. A questionnaire has been constructed for the patient groups in the study to register the clinical signs and symptoms. The patients will fill out the questionnaire before and after the treatment. The study patients will be followed up after treatment at the outpatient clinic at 1 and 3 months and at 1, 2, 5, and 10 years. Duplex ultrasound will be performed at all follow-up time points.

Furthermore, changes in the health-related quality of life (QoL) will be investigated in the study individuals. The EuroQol 5D (EQ5D) questionnaire will be used to assess the QoL of the study patients. The patients will fill out the EQ5D at inclusion in the study and 1, 2, 5, and 10 years after treatment of CMI and MALS in the patient groups. EQ-5D can be converted to a single summary index by applying a formula that attaches weight to each of the levels in each dimension. The EQ-5D index is varying between 0 to 1 where 1 presents best health condition and 0 presenting the worst health state .

Information from the quality of life and the costs of treatment during the hospital stay will be used to estimate the quality-adjusted life years (QALY) and the cost-utility of treating patients with CMI and MALS.

ELIGIBILITY:
Inclusion Criteria: Above 18 years and has given informed written consent for treatment and study participation

For the patient groups :

Group 1: Has CTA or ultrasound diagnosed MALS and is scheduled operative treatment.

Group 2: Has CTA or ultrasound diagnosed CMI and is scheduled operative or endovascular treatment.

For the control group:

Group 3- Has ultrasound based diagnosis of cholelithiasis and is scheduled for cholecystectomy.

Group 4- Has established Mb Crohn diagnosis and under gastric lab follow-up. Group 5- Young healthy blood donors of mean age 45 years and has excluded MALS or CMi with ultrasound.

Group 6- Healthy blood donors of mean age 70 years and has excluded MALS or CMi with ultrasound.

Exclusion Criteria: Age less than 18 years Has nor given written consent.

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: CMI and MALS patients with the vascular surgery department, Oslo University Hospital, with a consensus diagnosis of MALS and a diagnosis of CMI and schedules operative or endovascular treatment.
  Control groups are the individuals under treatment with the Oslo University Hospital or regular blood donors at the hospital.
Sampling Method: Non-Probability Sample
Enrollment: 180 (Estimated)
Dates: Start 2024-06-10 (Actual); Primary Completion 2037-05-31 (Estimated); Study Completion 2037-05-31 (Estimated)

PRIMARY OUTCOMES:
Plasma alpha Glutathione S transferase | 3 months
  This study compares the plasma Alpha GST in patients with CMI (n=30) and MALS (n=30) with those with 1-Morbus Crohn (n=30), 2-Gallstone disease (n=30), and age-matched healthy individuals (n=60).
  After inclusion in the study, blood tests will be performed to exclude renal failure and liver disease.
  Venous blood samples will be obtained before and 3 months after treatment in the patients with CMI and MALS. Blood samples will also be obtained from the individuals in the control groups twice ( at inclusion and 3 months apart ). The blood samples will be centrifuged and stored at -70 degrees until analyzed in batches with the ELISA technique.
  The plasma levels of Alpha GST in ng/mL before and after the intervention will be compared seperately for the differnt study groups.

SECONDARY OUTCOMES:
Health related quality of life (QoL) | 5 years
  Changes in the health-related quality of life (QoL) will be investigated. EuroQol 5D (EQ5D) questionnaire, which is a generic tool, will be used to assess the QoL of the study patients. EQ5D is a generic tool for the assessment of health related quality of life and is translated to Norwegian language and validated tool for the assessmeent of changes in the health related quality of life. The patients will fill out the EQ5D at inclusion in the study and 1, 2, 5, and 10 years after treatment of CMI and MALS in the patient groups. EQ5D has 5 questions with 5 levels of answers to each question. Level 1 will denote the best possible health status and level 5 denotes the worst health status for each of the 5 questions. It allows to a assess both physical and mental quality of health of the patients.
Clinical outcomes of the treatment of CMI and MALS | 10 years
  Effect of treatment on the symptoms of CMI and MALS postoperatively at 30 and 90 days, and at 1, 2, 5 and 10 years. A study specific questionnaire has been deveolped to register the signs and symptoms of CMI and MALS. The patients in the study will fill-out the questionnaire before and after the treatment and will repeat it at every follow-up time-point. The patients in the study will be follow-up by the clinicians who are not directly involved with the study and therefore the clinical information obtained will be standarized and made independent of the clinician's background. The questionnaire will allow to assess if the clinical symptoms have improved or worsen during the follow-up.
Cost utility analysis of the treatment of CMI and MALS | 5 years
  Quality adjusted life years (QALY ) estimation of the surgical and endovascular treatment of the patients with CMI and MALS. The costs of the treatment during the hospital stay will be calculated, compared with the costs of treatment given by the Norwegian Directorate of Health, QALY will be calculated based on the EQ5D results and the estimated treatment costs.
Intestinal ishemia biomarkers for CMI and MALS | 3 months
  Secondary outcome mesure: Plasma levels of intestinal fatty acid binding protein (iFABP) in ng/mL. In the previous studies, this biomarker has been demonstrated to be raised in the plasma of patients with CMI. Venous blood obtained fra the study individuals before and 3 months after the treatment of CMI and MALS will be analyzed with ELISA technique to discover any changes in these plasma biomarkers of ischemia. The groups will be compared for the changes in the individual plasma levels of these biomarkers and tested for any association to intestinal ischemia.
Plasma citruline | 3 months
  Plasma citroline is shown to be raised in the plasma of CMI patients in the previous studies. Venous blood samples will be taken before and 3 months after treatment of CMI and MALS patients and stored at -70 degrees until analyzed to find diffrences before and after the treatment and compare the diffrent study groups.
Immune modified albumin (IMA) | 3 months
  Immune modified albumin (IMA) in ng/mL is shown to be raised in the blood samples of patients with CMI. Venous blood samples will be taken before and 3 months after treatment of study patients with MALS, CMI and control groups. The blood samples will be analyzed to compare the plasma levels before and after the treatment of CMI and MALS and also compared with the control groups.

CONTACTS AND LOCATIONS:
Overall Officials: Syed Sajid Hussain Kazmi, MD, PhD, Principal Investigator — Department of vascular surgery, Oslo University Hospital
Locations (1):
- Department of vascular surgery, Oslo University Hospital, Oslo, Oslo County, Norway

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Kazmi SSH, Safi N, Berge ST, Kazmi M, Sundhagen JO, Julien K, Thorsby PM, Anonsen KV, Medhus AW, Hisdal J. Plasma alpha-Glutathione S-Transferase in Patients with Chronic Mesenteric Ischemia and Median Arcuate Ligament Syndrome. Vasc Health Risk Manag. 2022 Jul 21;18:567-574. doi: 10.2147/VHRM.S365625. eCollection 2022. PMID 35903288